CLINICAL TRIAL: NCT05055531
Title: "Effects of the Vaccin Against COVID 19 in a Cohort of Dialysis Patients: Adverse Events and Immunological Response"
Acronym: VACOVEIRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Raincy Montfermeil Hospital Group (Network)
Responsible Party: Sponsor
Other Study IDs: CHIM-GHT : RNI-3_02
Record Dates: First submitted 2021-09-17; First posted 2021-09-24 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-02

CONDITIONS: COVID Epidemic
Keywords: dialysis patients; vaccination; immunological response; mRNA vaccine; Vaccine safety; adverse event

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pandemic caused by COVID 19 continues to pose a threat to public health worldwide. Currently, approximately 2,397,312 people have died from it and 108,715,375 confirmed cases have been reported, according to the World Health Organization (WHO) as of February 13, 2021.

Patients with chronic kidney disease (CKD) are, from stage 3, at risk for a severe form of COVID 19 and this risk increases with the severity of the disease, including in dialysis or transplant patients according to the press release. HAS of December 2020.

As a result, France has prioritized vaccination for these patients the mRNA vaccine Therefore, the objective of this work is to study the safety of the vaccine in a population of hemodialysis patients in a heavy center, and the efficacy on the immune response (IgG) and the kinetics induced after 3 doses of the anti-Covid vaccine. to RNA.

DETAILED DESCRIPTION:
The pandemic caused by COVID 19 continues to pose a threat to public health worldwide. Currently, approximately 2,397,312 people have died from it and 108,715,375 confirmed cases have been reported, according to the World Health Organization (WHO) as of February 13, 2021.

Patients with chronic kidney disease (CKD) are, from stage 3, at risk for a severe form of COVID 19 and this risk increases with the severity of the disease, including in dialysis or transplant patients according to the press release. HAS of December 2020.

As a result, France has prioritized the mRNA vaccine vaccination for these patients in accordance with the vaccination strategy defined by the Minister of Health on Friday, January 15, 2021.

Phase 3 trials of RNA vaccines have shown good tolerability and greater than 90% efficacy in preventing symptomatic infection after two doses given 3 to 4 weeks apart , but hemodialysis patients did not not included in the first clinical trials of Covid-19 vaccination. Little is known about the immunological response to the COVID 19 vaccine, as is the need for new doses, given the usually low immune response in this population . Seroconversion after confirmed infection approaches 100% in the dialysis population, but the durability of this protective immune response remains uncertain. Some studies indicate that the IgG titers of COVID 19 decrease considerably after 3 months Therefore, the objective of this work is to study the safety of the vaccine in a population of hemodialysis patients in a heavy center, and the efficacy on the immune response (IgG) and the kinetics induced after 3 doses of the anti-Covid vaccine. All patients at the dialysis center were offered the coronavirus vaccine. The vaccination was carried out during a dialysis session. The vaccines administered were the only ones to have had Marketing Authorization from January 2021: Pfizer / BioNTech and Moderna. Not all patients were vaccinated at the same time. The first doses given to the first dialysis patients were given in January 2021, then the injections were staggered over time. In accordance with the recommendations of the Ministry of Health, patients were offered 3 doses of vaccine (from the same laboratory).

ELIGIBILITY:
Inclusion Criteria:

* Chronic prevalent hemodialysis patients (for more than 3 months) performing 2 to 3 sessions / week, at least 3 hours, at the André Grégoire hospital center, Montreuil.
* Age> 18 years old,
* Vaccination of at least one dose of Pfizer or Moderna vaccine from January 1, 2021, performed during a dialysis session.
* Affiliation to a social security scheme;

Exclusion Criteria:

* Acute hemodialysis (duration <3 months).
* Patient who died before the first vaccine dose.
* Age <18 years old
* Inability to give consent (eg mental retardation, patient under guardianship or legal protection, decompensated psychiatric illness, too advanced dementia (MMS <15/30, etc.)
* Pregnant women
* Patient participating in another interventional study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease (CKD) are, from stage 3, or a population of hemodialysis patients at risk of severe form of COVID 19
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-08 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Vaccine safety | 6 months
  number of clinical adverse events and consequences on dialysis treatment related to vaccination against SARS COV 2

SECONDARY OUTCOMES:
the immunological response | 6 months
  he immunological response by assaying the IgGs of dialysis patients from the second vaccine dose and in the 6 months that follow.

CONTACTS AND LOCATIONS:
Locations (1):
- GAUTHIER, Montreuil, France

IPD SHARING:
Plan to Share IPD: No